CLINICAL TRIAL: NCT01407133
Title: Assessment of Conventional Repetitive Transcranial Magnetic Stimulation for the Treatment of Chronic Tinnitus
Brief Title: Conventional Repetitive Transcranial Magnetic Stimulation for Tinnitus Treatment
Acronym: MagTIN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2004.365
Record Dates: First submitted 2011-07-26; First posted 2011-08-02 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Chronic Tinnitus
Keywords: Neuro-otology; Chronic tinnitus; Sensory disability; Repetitive transcranial magnetic stimulation; Dose escalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active rTMS (Experimental): 48 subjects will receive active temporal rTMS, applied with the following combined parameters:
  * intensity: 100% of resting motor threshold
  * stimulation frequency: low-frequency continuous stimulation (0.5 or 1 Hz) or high-frequency stimulation trains (4 or 12 Hz)
  * number of stimulations per session: 300, 900 or 1800 per session
  * number of sessions per week: spaced out / low density protocol (1 per week) or dense / high density protocol (5 per week)
  * total number of sessions for the whole intervention: short protocol (5 sessions) or long protocol (20 sessions).
  Interventions: Device: transcranial magnetic stimulator (class 2b) Medtronic © MagPro X100 (with MagOption) stimulator and Butterfly Coil MCF-B65 (figure-8 coil with fluid cooling)
- Sham rTMS (Sham Comparator): 16 subjects will receive sham rTMS, applied with the same combination of parameters as active rTMS, except for the number of stimulations per session (300 or 900)
  Interventions: Device: Sham transcranial magnetic stimulator Medtronic © MagPro X100 (shielded figure-8 coil with fluid cooling)

INTERVENTIONS:
Device: transcranial magnetic stimulator (class 2b) Medtronic © MagPro X100 (with MagOption) stimulator and Butterfly Coil MCF-B65 (figure-8 coil with fluid cooling) — The study is based on a dual procedure consisting of comparisons between active and sham rTMS on the one hand and between four increasing levels of magnetic "pseudo-dose" on the other hand. Each level comprises 16 patients randomly assigned to active rTMS group (12 patients) or sham rTMS group (4 patients). The transition from one level to another is authorized by an independent oversight committee charged with checking the tolerability of rTMS sessions for the tested level. The neuronavigated rTMS use either active or sham figure-eight coil and is centered over the primary auditory cortex contralateral to the perceived predominant side of tinnitus. This target is located through anatomical brain MRI and neuronavigated brain system. According to the stimulation parameters, each rTMS session can last from 5 to 112 minutes and the whole rTMS intervention from 1 to 20 weeks. The follow-up is spread over twelve months.
  Other Names: Medtronic © MagPro X100 (with MagOption) stimulator and Butterfly Coil MCF-B65 (figure-8 coil with fluid cooling)
  Arms: Active rTMS
Device: Sham transcranial magnetic stimulator Medtronic © MagPro X100 (shielded figure-8 coil with fluid cooling) — Same sound level as active rTMS, but magnetic field strongly attenuated
  Other Names: Medtronic © MagPro X100 (with MagOption) stimulator and Placebo Butterfly Coil MCF-P-B65 (shielded figure-8 coil with fluid cooling)
  Arms: Sham rTMS

SUMMARY:
The objective of the investigators study is to assess conventional repetitive transcranial magnetic stimulation (rTMS) in patients with chronic severe tinnitus. A randomized, double-blind, sham-controlled procedure, with four increasing levels of magnetic "pseudo-dose" has been designed, in order to characterize the effectiveness of rTMS while controlling its safety and tolerability. By combining various rTMS protocols with a twelve-month follow-up, and using an effect modeling, the study aims at: (i) specify the effective values of rTMS parameters, with an adequate tolerance; (ii) determine the expected benefit and the persistence of effect; (iii) assess the practical feasibility of this kind of therapeutic management.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 75 years old;
* Adequate medical condition (ASA P1 or P2 in Physical Status Classification System);
* Disabling tinnitus (STSS > 8/16 or THQ > 50%), with the following characteristics: continuous, subjective, non-pulsatile; unilateral (or bilateral with unilateral predominance), chronic (duration for at least one year), refractory for usual treatments taken for at least six months;
* Naive regarding TMS;
* Able to provide informed consent.

Exclusion Criteria:

* Objective tinnitus or tinnitus with treatable cause;
* Presence of intracranial or intraocular ferromagnetic materiel or particles (with the exception of dental fillings and MRI-compatible stapedectomy prosthesis);
* Cardiac pacemaker or other electronic implants (including cochlear implant);
* Serious heart disease or other unstable major medical condition;
* Personal history of central nervous system disorder, head injury, stroke or seizures (including childhood febrile seizures);
* Familial history of epilepsy;
* Concomitant medication with antidepressants and antipsychotics;
* Possibility of pregnancy;
* Known claustrophobia;
* Others known contraindications to rTMS or brain MRI;
* Refusal to be informed about the results of anatomical MRI

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in tinnitus perception, as measured over time using a visual analog rating scale (subjective loudness of tinnitus) | At subject enrollment; daily for 2 weeks before the intervention; before and after each rTMS session, once at the end of each week and at the end of intervention; during follow-up: twice a week for 6 months, and 1 year after the end of intervention
  The time between enrollment and rTMS intervention will vary from one subject to another (expected average of 4 months); depending on the protocol, the end of the intervention corresponds to the end of week 1, 4, 5 or 20 (first day of rTMS as reference)

SECONDARY OUTCOMES:
Tolerance of rTMS, evaluated through a semi-structured interview on specific and nonspecific adverse events | After the first rTMS session; before and after each following session and at the end of intervention period; 1, 4 or 5, and 20 weeks after the start of intervention; 1, 3, 6 months and 1 year after the end of intervention
  Depending on the protocol, the end of the intervention corresponds to the end of week 1, 4, 5 or 20 (first day of rTMS as reference)
Auditory status, evaluated through tonal audiometry (pure-tone average) | At subject enrollment; before the first rTMS session and after the last rTMS session (for all types of protocols), and every five sessions of rTMS (for long protocols)
  The time between enrollment and rTMS intervention will vary from one subject to another (expected average of 4 months)
Change in severity of tinnitus, measured through a multidimensional self-questionnaire: Subjective Tinnitus Severity Scale (STSS) | At subject enrollment; before the first rTMS session, in the middle and at the end of intervention period; 1, 4 or 5, and 20 weeks after the start of intervention; 1, 3, 6 months and 1 year after the end of intervention
  Depending on the protocol, middle (respectively, end) of the intervention corresponds to day 3, day 12, beginning of week 3 or beginning of week 11 (respectively, end of week 1, 4, 5 or 20), with the first day of rTMS as reference
Change in handicap related to tinnitus, measured through a multidimensional self-questionnaire: Tinnitus Handicap Questionnaire (THQ) | At subject enrollment; at the beginning, in the middle and at the end of rTMS intervention period; 1, 4 or 5, and 20 weeks after the start of intervention; 1, 3, 6 months and 1 year after the end of intervention
Change in hyperacusis, measured through a multidimensional self-questionnaire: Auditory Hypersensitivity Questionnaire | At subject enrollment; at the beginning, in the middle and at the end of rTMS intervention period; 1, 4 or 5, and 20 weeks after the start of intervention; 1, 3, 6 months and 1 year after the end of intervention
Change in anxiety and depression, measured through a two-dimensional self-questionnaire: Hospital Anxiety and Depression Scale (HADS) | At subject enrollment; at the beginning, in the middle and at the end of rTMS intervention period; 1, 4 or 5, and 20 weeks after the start of intervention; 1, 3, 6 months and 1 year after the end of intervention
Personality, assessed through a multidimensional self-questionnaire: Mini-Mult (short form of the MMPI) | At subject enrollment
  The time between enrollment and rTMS intervention will vary from one subject to another (expected average of 4 months)
Change in tinnitus spectrum (loudness and pitch), characterized through psychoacoustical measurements: tinnitometry | At subject enrollment; at the beginning, in the middle and at the end of rTMS intervention period; 1, 4 or 5, and 20 weeks after the start of intervention; 1, 3, 6 months and 1 year after the end of intervention
Motivation level, assessed through a short self-questionnaire (Likert-type scale) | At the beginning of intervention period (before the first rTMS session) (day 1)
Satisfaction degree, assessed through a short self-questionnaire (Likert-type scale) Time Frame: At the end of SMTr intervention | At the end of intervention period (end of week 1, 4, 5 or 20, with the first day of rTMS as reference)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier PERROT, MD, PhD, Principal Investigator — Service d'Audiologie et Explorations Orofaciales (Pr. COLLET) - Centre Hospitalier Lyon Sud - Hospices Civils de Lyon
Locations (3):
- France (3):
  - Département d'ORL et de Chirurgie Cervico-Maxillo-Faciale, Hôpital Edouard Herriot, Lyon
  - Service d'Audiologie et Explorations Orofaciales, Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Service d'Oto-Rhino-Laryngologie, Centre Hospitalier Lyon-Sud, Pierre-Bénite

REFERENCES:
- [Result] Tringali S, Perrot X, Collet L, Moulin A. Repetitive transcranial magnetic stimulation (rTMS) noise: a relevance for tinnitus treatment? Brain Stimul. 2012 Oct;5(4):655-6. doi: 10.1016/j.brs.2011.10.006. Epub 2012 Feb 22. No abstract available. PMID 22405743
- [Result] Tringali S, Perrot X, Collet L, Moulin A. Repetitive transcranial magnetic stimulation noise levels: methodological implications for tinnitus treatment. Otol Neurotol. 2012 Sep;33(7):1156-60. doi: 10.1097/MAO.0b013e318263d37d. PMID 22872177
- [Result] Tringali S, Perrot X, Collet L, Moulin A. Repetitive transcranial magnetic stimulation: hearing safety considerations. Brain Stimul. 2012 Jul;5(3):354-363. doi: 10.1016/j.brs.2011.06.005. Epub 2011 Jul 26. PMID 21824837